CLINICAL TRIAL: NCT02049749
Title: Improving Child Behavior Problems in the Primary Care Setting
Brief Title: Parent Program to Improve Child Behavior Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 13-010728
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-01

CONDITIONS: Child Behavior Problems
Keywords: Child Behavior Problems; Parent Training Program

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed CARE (No Intervention): 40 child-caregiver pairs will be randomized to usual treatment plus delayed CARE (control). Under usual treatment, patients will be referred to a behavioral health specialist at the discretion of their pediatrician and the office social worker for additional diagnosis and treatment and/or provided with a 1-2 page informational handout on child behavior problems from the CHOP patient care manual. Following the final interview (3-4 months after enrollment for each subject) all participants randomized to the control arm (usual treatment plus delayed CARE) will receive the CARE training, if desired.
- Immediate CARE (Experimental): 40 child-caregiver pairs will be randomized to usual treatment plus immediate CARE. The trainings are administered to groups of 4-10 caregivers at a time and are led by two mental health providers trained in the CARE curriculum. The children do not attend the training; however, caregivers are expected to practice the skills that they learn in CARE with their child between sessions. The curriculum involves 6 sessions over 6-8 weeks. Each session will be 1-2 hours.
  Interventions: Behavioral: Immediate CARE

INTERVENTIONS:
Behavioral: Immediate CARE — CARE is a group parent training informed by the principles of Parent Child Interaction Therapy and was developed by Trauma Treatment Training Center and CHOP Policy Lab. CARE has been used in many populations including residential treatment center/domestic violence shelter staff, daycare providers, graduate students, biological parents, and foster parents/caseworkers. Goals are to decrease stress for caregivers, improve child behavior, and enhance the caregiver-child relationship, family stability, and wellness. The training teaches parents to follow a child's lead thus building a connection and promoting positive behaviors. The focus is on giving attention to child's pro-social behavior and ignoring minor misbehavior. The second phase teaches techniques for giving effective commands.
  Other Names: Child Adult Relationship Enhancement (CARE)
  Arms: Immediate CARE

SUMMARY:
The purpose of this research study is to learn whether or not a brief parenting program called Child Adult Relationship Enhancement (CARE) offered at a primary care office can help improve behavior problems in children who are 2-6 years old.

DETAILED DESCRIPTION:
The study will be a randomized controlled trial (RCT) of the CARE intervention. The study will include 2-6 year old children who receive their primary care at the Children's Hospital of Philadelphia, South Philadelphia Primary Care clinic and whose caregiver and/or doctor has concern about a behavior problem in the child. The caregivers will also be subjects in the study.

Child-caregiver pairs who agree to be in the study will be randomly assigned to receive the CARE training immediately or in 3-4 months.

The CARE intervention will last 6 weeks and child behavior and parenting will be measured at baseline, 6-8 weeks, and 14-18 weeks. Investigators will also measure parent satisfaction with the CARE intervention.

* Child Adult Relationship Enhancement (CARE) is a group parent training program.
* The goals of the program are to teach parents skills that help their children successfully reach developmental milestones while increasing positive behaviors.
* The program also was designed to help parents manage and decrease negative child behaviors.
* Each training will be led by 2 therapists and 4-10 parents will attend the CARE program together.
* Children do not attend the training but parents are encouraged to practice the skills learned at CARE between the sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Caregiver is 18 years or older
2. Caregiver is English speaking
3. Child is 2-6 years old
4. Caregiver reports that child has a behavior problem
5. Child attends CHOP South Philadelphia Primary Care for primary care
6. Parental/guardian permission is provided (informed consent)

Exclusion Criteria:

1. Child has a cognitive age less than 2 years old as determined by the referring clinician
2. Child is already receiving behavioral health therapy or medication (other than medication for Attention Deficit Hyperactivity Disorder)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-05; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne N Wood, MD, MSHP, Principal Investigator — CHOP
Locations (1):
- CHOP Primary Care, South Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- No Intervention: Delayed CARE: 40 child-caregiver pairs will be randomized to usual treatment plus delayed PriCARE (control). Under usual treatment, patients will be referred to a behavioral health specialist at the discretion of their pediatrician and the office social worker for additional diagnosis and treatment and/or provided with a 1-2 page informational handout on child behavior problems from the CHOP patient care manual. Following the final interview (3-4 months after enrollment for each subject) all participants randomized to the control arm (usual treatment plus delayed PriCARE) will receive the PriCARE training, if desired.
- Experimental: Immediate CARE: 80 child-caregiver pairs will be randomized to usual treatment plus immediate PriCARE, a 6 session adaptation of the CARE group parent training. CARE was developed by Trauma Treatment Training Center and informed by the principles of Parent Child Interaction Therapy. CARE has been used in many populations including daycare providers, biological parents, and foster parents. Goals are to decrease caregiver stress, improve child behavior, and enhance the caregiver-child relationship, family stability, and wellness. CARE teaches parents to follow a child's lead thus building a connection and promoting positive behaviors. CARE focuses on giving attention to child's pro-social behavior and ignoring minor misbehavior. CARE teaches techniques for giving effective commands. The PriCARE curriculum involves 6 1-2 hour sessions over 6-8 weeks. 2 mental health providers lead PriCARE trainings for groups of 4-10 caregivers. Children do not attend PriCARE.
Period: Overall Study
Arm/Group | No Intervention: Delayed CARE | Experimental: Immediate CARE
Started | 80 (40 children plus 40 caregivers) | 160 (80 children plus 80 caregivers)
Completed | 80 | 160 (80 children plus 80 caregivers)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experiemental: Immediate CARE: 80 child-caregiver pairs will be randomized to usual treatment plus immediate PriCARE, a 6 session adaptation of the CARE group parent training. CARE was developed by Trauma Treatment Training Center and informed by the principles of Parent Child Interaction Therapy. CARE has been used in many populations including daycare providers, biological parents, and foster parents. Goals are to decrease caregiver stress, improve child behavior, and enhance the caregiver-child relationship, family stability, and wellness. CARE teaches parents to follow a child's lead thus building a connection and promoting positive behaviors. CARE focuses on giving attention to child's pro-social behavior and ignoring minor misbehavior. CARE teaches techniques for giving effective commands. The PriCARE curriculum involves 6 1-2 hour sessions over 6-8 weeks. 2 mental health providers lead PriCARE trainings for groups of 4-10 caregivers. Children do not attend PriCARE.
- Total: Total of all reporting groups
Arm/Group | No Intervention: Delayed CARE | Experiemental: Immediate CARE | Total
Number analyzed (Participants) | 80 | 160 | 240
Age, Categorical [Count of Participants; unit: Participants] — For child participants age in years was collected. For caregiver participants age was categorized as 18-29 years, 30-39 years, or 40-49 years, 50-59 years, 60-69 years, or 70 plus years. There were 3 caregivers in the 60-69 years for which it is unknown whether they were <65 or >65. For reporting purposes these 3 caregivers are included in the < 65 category in the table below.
  Participants
    <=18 years | 40 | 80 | 120
    Between 18 and 65 years | 40 | 80 | 120
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 105 | 163
  Male | 22 | 55 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 22 | 33
  Not Hispanic or Latino | 68 | 138 | 206
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 54 | 103 | 157
  White | 22 | 46 | 68
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 5 | 5
Caregiver relationship to child [Count of Participants; unit: Participants] — Population: Caregiver relationship is provided for caregiver participants only
  Participants
    number analyzed (Participants) | 40 | 80 | 120
    Mother | 40 | 74 | 114
    Father | 0 | 1 | 1
    Grandmother | 0 | 5 | 5
ECBI Problem Scale [Mean (Standard Deviation); unit: units on a scale] — The Eyberg Child Behavior Inventory (ECBI) is a 36 item parent rating scale that measures problem behaviors (externalizing or conduct-disordered behaviors) in children 2-16 on the Intensity scale and the Problem scale. The problem score (range 0-36) is the total number of behaviors for which the parent identifies that the behavior is problematic. Higher scores indicate worse behavioral problems. Baseline ECBI Problem Scale was collected by parental report for Child Participants only. Population: ECBI measures were only collected on child participants and not caregivers
  units on a scale
    number analyzed (Participants) | 40 | 80 | 120
    (all) | 18 (8) | 21 (8) | 20 (8)
ECBI Intensity Scale [Mean (Standard Deviation); unit: units on a scale] — The Eyberg Child Behavior Inventory (ECBI) is a 36 item parent rating scale that measures problem behaviors (externalizing or conduct-disordered behaviors) in children 2-16 on the Intensity scale and the Problem scale. Each of the 36 behaviors is rated on a 7-point intensity scale. The Intensity score (range 36-252) is the total frequency of occurrence for the behaviors. Higher scores indicate worse behavioral problems. Baseline ECBI Intensity Scale was collected by parental report for Child Participants only. Population: ECBI Measures only collected for child participants.
  units on a scale
    number analyzed (Participants) | 40 | 80 | 120
    (all) | 139 (39) | 153 (39) | 149 (40)
Adult Adolescent Parenting Inventory 2 (AAPI2) [Mean (Standard Deviation); unit: units on a scale] — Adult Adolescent Parenting Inventory 2 (AAPI-2) is a 40-item parent self-report measure that assesses parenting attitudes on five subscales: 1) inappropriate expectations of children 2) parental lack of empathy towards child's needs, 3) strong belief in the use of corporal punishment as a means of discipline, 4) reversing parent-child role responsibilities and 5) oppressing child's power and independence. Standardized sten scores for each of the 5 subscales range from 1-10 with lower scores indicating higher risk for child maltreatment. Population: AAPI scores were only measured and reported for caregiver participants
  units on a scale
    Expectations: number analyzed (Participants) | 40 | 80 | 120
    Expectations | 4.45 (1.53) | 4.66 (1.66) | 4.59 (1.62)
    Empathy: number analyzed (Participants) | 40 | 80 | 120
    Empathy | 4.23 (2.14) | 4.21 (2.06) | 4.22 (2.08)
    Corporal Punishment: number analyzed (Participants) | 40 | 80 | 120
    Corporal Punishment | 5.40 (1.37) | 5.67 (1.78) | 5.58 (1.66)
    Parent-child roles: number analyzed (Participants) | 40 | 80 | 120
    Parent-child roles | 5.30 (2.14) | 5.16 (2.32) | 5.21 (2.26)
    Power and independence: number analyzed (Participants) | 40 | 80 | 120
    Power and independence | 5.22 (2.12) | 5.20 (1.93) | 5.21 (1.99)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Eyberg Child Behavior Inventory (ECBI) Score at Different Time Points (Baseline up to 18 Weeks)
Description: Behavior will be measured by the Eyberg Child Behavior Inventory (ECBI). The primary outcome is the ECBI change score (time 3-time1). The ECBI is a parent rating scale designed to measure conduct problem behaviors in children ages 2-16 years. The instrument contains 36 items that assess behavior on two scales. The problem scale provides a yes/no problem identification rating for each item, and the sum of yes responses yields a problem score with a potential range from 0 to 36 with a clinical cutoff of 15. The intensity scale provides a frequency-of-occurrence rating for each item, ranging from never (1) to always (7) and the ratings are summed to yield an intensity score with a potential range from 36 to 252 with a clinical cutoff of 131. Higher scores indicate worse outcomes. The ECBI has demonstrated strong internal consistency, test-retest reliability, and discriminant validity and has been shown to be a sensitive indicator of intervention efficacy for child behavior problems.
Time Frame: Mean Change in ECBI Scores from Baseline to 14-18 weeks. Decreases in ECBI scores reflect improvements in behavior.
Population: Eyberg Child Behavior Inventory (ECBI) is a 36 item parent rating scale that measures problem behaviors in children 2-16 on the problem scale and intensity scale.The intensity score (range 36-252) is the total frequency of occurrence for the behaviors. The problem score (range 0-36) is the total number of behaviors for which the response is "yes".
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | No Intervention: Delayed CARE | Experiemental: Immediate CARE
Number analyzed (Participants) | 40 | 80
units on a scale
  Adjusted ECBI Intenstity Change Score | -7 [-17 to 2] | -22 [-29 to -16]
  Adjusted ECBI Problem Change Score | -2 [-4 to 0] | -5 [-7 to -4]

2. Secondary Outcome: Changes From Baseline in Parental Disciplinary Practices Assessed at Different Time Points (Baseline up to 18 Weeks)
Description: Investigators want to determine the effect of the CARE intervention on diminishing harsh parenting as measured by the Adult Adolescent Parenting Inventory-2.
  The Adult Adolescent Parenting Inventory-2 (AAPI-2) is a 40 item parent-report measure that assesses parenting attitudes along 5 dimensions: inappropriate expectations of children, parental lack of empathy towards children's needs, strong belief in the use of corporal punishment as a means of discipline, reversing parent-child role responsibilities, and oppressing children's power and independence.
  Parents respond to each item on a five point Likert Scale of Strongly Agree, Agree, Disagree, Strongly Disagree and Uncertain. This measure yields a score of 1-10 for each construct. Higher scores indicate lower risk parenting.
Time Frame: Mean change in scores from baseline to 14-18 weeks. Increases in scores indicate decreased risk for abuse and better outcomes.
Population: Adult Adolescent Parenting Inventory (AAPI-2): assesses 5 parenting constructs:1) inappropriate expectations of child,2) lack of empathy towards child's needs,3)belief in corporal punishment, 4) reverses parent-child roles, 5) restricts child's power and independence.Range for each scale is 1-10. Lower numbers indicate higher abuse risk.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Intervention: Delayed CARE | Experimental: Immediate CARE
Number analyzed (Participants) | 40 | 80
units on a scale
  Expectations of Children | 0.575 (1.56) | 0.362 (1.46)
  Parental Empathy toward Children's Needs | 0.25 (1.58) | 0.825 (1.57)
  Use of Corporal Punishment | -0.25 (1.19) | 0.2 (1.03)
  Parent-Child Family Roles | 0.425 (1.29) | 0.875 (1.79)
  Children's Power and Independence | -0.65 (2.15) | 0.375 (1.84)

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- No Intervention: Delayed CARE: 40 child-caregiver pairs will be randomized to usual treatment plus delayed CARE (control). Under usual treatment, patients will be referred to a behavioral health specialist at the discretion of their pediatrician and the office social worker for additional diagnosis and treatment and/or provided with a 1-2 page informational handout on child behavior problems from the CHOP patient care manual. Following the final interview (3-4 months after enrollment for each subject) all participants randomized to the control arm (usual treatment plus delayed CARE) will receive the CARE training, if desired.
- Experiemental: Immediate CARE: 80 child-caregiver pairs will be randomized to immediate CARE. Immediate CARE: CARE is a group parent training informed by the principles of Parent Child Interaction Therapy and was developed by Trauma Treatment Training Center and CHOP Policy Lab. CARE has been used in many populations including residential treatment center/domestic violence shelter staff, daycare providers, graduate students, biological parents, and foster parents/caseworkers. Goals are to decrease stress for caregivers, improve child behavior, and enhance the caregiver-child relationship, family stability, and wellness. The training teaches parents to follow a child's lead thus building a connection and promoting positive behaviors. The focus is on giving attention to child's pro-social behavior and ignoring minor misbehavior. The second phase teaches techniques for giving effective commands.
Arm/Group | No Intervention: Delayed CARE | Experiemental: Immediate CARE
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/160
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/160
Other Adverse Events (participants affected / at risk) | 0/80 | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No